CLINICAL TRIAL: NCT04293237
Title: Metric Charcteristics of Sit-to-stand Tests in Patients After Lower-limb Amputation
Acronym: STST
Status: Completed | Type: Observational
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Responsible Party: Sponsor
Other Study IDs: URIS202002
Record Dates: First submitted 2020-02-26; First posted 2020-03-03 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Lower Limb Amputation
Keywords: unilateral lower-limb amputation; sit-to-stand tests; walking tests; psychometric characteristics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to assess various aspects of reliability and validity of two sit-to-stand tests, the Five Times Sit to Stand Test (5TSTS) and the 30-Second Sit to Stand Test (30SSTS). The tests will be performed by patients after lower-limb amputation who have been newly fitted with a prosthesis. Each test will be performed with and without the prosthesis on two occasions: on the first day when the patients will be able to walk independently with their prosthesis and two weeks later. On the same two occasions, the patients will also perform three walking tests (in randomised order): the L-test, the 10-Metre Walk Test and the 6-Minute Walk Test. In addition, the patients will repeat the 5TSTS and the 30SSTS one day after the first assessment. The results will be used to detect the presence of a floor effect, assess repeatability and concurrent validity, as well as estimate minimal detectable change and effects size for the effect of rehabilitation.

DETAILED DESCRIPTION:
All the tests will be performed using standardised protocols and technical aids. The assessments will be performed in the afternoon (after the daily rehabilitation program). The patients who will be able to perform the 5TSTS will perform that test first. If those patients will bill able to stand up within 30 seconds on each of the five trials, the 30SSTS will be performed next; otherwise, the number of times that the patient was able to complete the transition to the standing position will be recorded and taken as the 30SSTS result. Repetition of the outcome measurements will not serve to simply use the differences as the actual outcomes, but will serve to assess floor effect (the percentage of patients attaining the minimum possible score) on each occasion, to assess repeatability (intra-class correlation between the measurements on two consecutive days), minimal detectable change (calculated from the standard error of measurement, which will be estimated from the correlation between the measurements at the start and after two weeks) and effect size (difference between the mean measurements at the start and after two weeks, divided by the standard deviation at the start). In addition, the repeated measurements will be used to assess concurrent validity in terms of the correlation between the sit-to-stand tests and the walking tests on two occasions (at the start and after two weeks).

ELIGIBILITY:
Inclusion Criteria:

* unilateral trans-femoral or trans-tibial amputation
* fitted with a prosthesis for the first time
* being able to walk with the prosthesis independently (without walking aids or using a cane, crutch or walker)

Exclusion Criteria:

* balance disorder beacuse of neurological disease
* other muskuloskeletal impairments affecting the outcome measurements
* cardio-vascular disease that could be worsened by prforming the outcome measurements
* general ill health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to impatient rehabilitation at the Department for Rehabilitation of Patients after Amputation of the University Rehabilitation Institute in Ljubljana, Slovenia, who will meet the inclusion criteria and not meet any of the exclusion criteria will be consecutively recruited until the planned sample size is reached
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2020-05-09 (Actual); Study Completion 2020-05-09 (Actual)

PRIMARY OUTCOMES:
Five Times Sit to Stand Test (5TSTS) - Start | At the start of the study
  The 5TSTS assesses functional lower extremity strength, transitional movements and balance. The outcome is the tame required by the participant to complete the task.
Five Times Sit to Stand Test (5TSTS) - After one day | One day after the start of the study
  The 5TSTS assesses functional lower extremity strength, transitional movements and balance. The outcome is the tame required by the participant to complete the task.
Five Times Sit to Stand Test (5TSTS) - After two weeks | Two weeks after the start of the study
  The 5TSTS assesses functional lower extremity strength, transitional movements and balance. The outcome is the tame required by the participant to complete the task.
30-Second Sit to Stand Test (30SSTS) - Start | At the start of the study
  The 30SSTS assesses leg strength and endurance. The outcome is the number of times that the participant is able to completely stand up from the chair within 30 secons.
30-Second Sit to Stand Test (30SSTS) - After one day | One day after the start of the study
  The 30SSTS assesses leg strength and endurance. The outcome is the number of times that the participant is able to completely stand up from the chair within 30 secons.
30-Second Sit to Stand Test (30SSTS) - After two weeks | Two weeks after the start of the study
  The 30SSTS assesses leg strength and endurance. The outcome is the number of times that the participant is able to completely stand up from the chair within 30 secons.

SECONDARY OUTCOMES:
L-test | At the start of the study and after two weeks
  The L-test is a performance-based measure of functional mobility. It is a modification of the Timed Up and Go test that overcomes the ceiling effect in higher-functioning patients. The participant must stand up from the chair, walk 7 m, turn 90 degrees, walk 3 m, then turn 180 degrees, and return along the same path to sit in the chair.
10-Metre Walk Test (10mWT) | At the start of the study and after two weeks
  The 10mWT assesses walking speed over a short duration.
6-Minute Walk Test (6mWT) | At the start of the study and after two weeks
  The 6mWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Podlogar, MPT, Principal Investigator — University Rehabilitation Institute, Republic of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No